CLINICAL TRIAL: NCT05591820
Title: A Randomized Controlled Trial on Brief Behavioral Parent Training Versus Care as Usual in Children With Behavioral Difficulties
Brief Title: A Randomized Controlled Trial on Brief Behavioral Parent Training
Acronym: PAINT-GGZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METc 2022/221; file number 60-63600-98-1 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Disruptive Behavior; Behavior Problems; Behavioral Problems; Problem Behaviors; Behavioral Symptoms; Behavioral Difficulties
Keywords: Parent Training; Behavioral Parent Training; Brief Parent Training; Individually-Tailored Parent Training; Booster Sessions; Disruptive Behavior; Children; Randomized Controlled Trial; Clinical Trial; Brief Treatment
MeSH Terms: conditions — Problem Behavior; Mental Disorders; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: To examine the research objectives, a randomized controlled trial with two arms is used. Referred children and their parents will be randomly assigned (equal randomization) to (a) brief parent training, with optional booster sessions up to one year after the training, or (b) care as usual (CAU), as regularly provided by the mental health centers involved. Children in the brief parent training group will not receive CAU until the first posttreatment assessment (T1). After that, CAU is allowed and parents can make use of booster sessions (maximum once every four weeks) with the therapist who provided the training.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors who will code the records of mealtime routines made by parents will be unaware of in which arm parents in the study are participating. The audio records will therefore be a masked measure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief behavioral parent training with optional booster sessions (Experimental): A brief, individualized, three-session parent training that exists of two (bi)weekly individually tailored training sessions of two hours and a third session of one hour in which the training will be evaluated, and maintenance training will be provided. After that, parents wishing to receive additional support can receive single booster sessions maximum once every four weeks and/or receive care as usual.
  Interventions: Behavioral: Brief behavioral parent training with optional booster sessions
- Care as usual (CAU) (Active Comparator): The care that is usually provided by the clinical institutions to treat children's disruptive behaviors. There will be no restrictions regarding type or duration of CAU (only the brief parent training will not be allowed) which may for example include psychoeducation, (long) parent training, child treatment (e.g., pharmacotherapy, cognitive behavioral therapy) or family therapy.
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Brief behavioral parent training with optional booster sessions — A brief and individually-tailored behavioral parent training program that combines stimulus control and contingency management techniques to treat children's behavioral difficulties in three (bi)weekly sessions and optional booster sessions.
  Other Names: PAINT-P (Parent); PAINT-GGZ; Brief parent training
  Arms: Brief behavioral parent training with optional booster sessions
Behavioral: Care as usual — The care that is usually provided by the clinical institutions to treat children's behavioral difficulties. There are no restrictions regarding type or duration of CAU (only the brief parent training will not be allowed) which may for example include psychoeducation, (long) parent training, child treatment (e.g., pharmacotherapy, cognitive behavioral therapy) or family therapy.
  Other Names: CAU
  Arms: Care as usual (CAU)

SUMMARY:
RATIONALE: The access to and uptake of evidence-based behavioral parent training for children with behavioral difficulties (i.e., oppositional, defiant, aggressive, hyperactive, impulsive, and inattentive behavior) are currently limited because of a scarcity of certified therapists and long waiting lists. These problems are in part due to the long and sometimes perceived as rigid nature of most evidence-based programs and result in few families starting behavioral parent training and high dropout rates. Brief and individually tailored parenting interventions may reduce these problems and make behavioral parent training more accessible.

OBJECTIVES: This project aims to increase the effective use of parent training for children with behavioral difficulties by (1) examining short and longer-term effectiveness of a new, brief, individual, and individually-tailored parent training program with optional booster sessions to prevent relapse, compared to care as usual (CAU); (2) assessing the cost-effectiveness of the brief parent training program compared to CAU.

STUDY DESIGN: In this two-arm, multi-center randomized controlled trial (RCT), parents are randomly assigned (1:1 ratio) to either (a) three sessions of brief behavioral parent training with optional booster sessions, or (b) CAU, as regularly provided by the involved mental healthcare centers. The study outcomes are measured at baseline before randomization (T0), one week after the third session for parents in the brief behavioral parent training arm and eight weeks after T0 for parents in the CAU arm (first posttreatment measurement, T1), six months after T1 (second posttreatment measurement, T2) and twelve months after T1 (third posttreatment measurement, T3).

STUDY POPULATION: Parents of children who experience behavioral difficulties in the home setting and were referred to a child mental healthcare center.

INTERVENTION: Parents in the intervention arm receive a short, individualized, three-session training primarily aimed at reducing children's behavioral problems. It exists of two (bi)weekly individually tailored training sessions of two hours and a third session of one hour in which the training will be evaluated, and maintenance training will be provided. After that, parents wishing to receive additional support can receive single booster sessions maximum once every four weeks and/or receive care as usual. Parents in the control arm receive care as usual for children's behavioral problems. The treatments in both arms are fully embedded in Dutch routine mental health care.

MAIN STUDY PARAMETERS: The primary outcome is the severity of four individual target behavioral difficulties that parents want to address in the training. Secondary outcomes are parent-reported behavioral difficulties, parent-reported child well-being, parent-reported parenting behaviors, masked audio records of mealtime routines to measure parent and child behavior, parent-reported parenting stress, parent-reported parenting self-efficacy, parent-reported parental attitude towards their child, consumption and cost of mental health care, and health state utility values. We furthermore measure evaluations of the program by parents and therapists and explore whether parental attachment, parental psychopathology, parental reward responsivity, parent-reported child reward responsivity and punishment sensitivity moderate the intervention effects.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   Behavioral difficulties, including oppositional, defiant, aggressive, hyperactive, impulsive, and inattentive behavior, are one of the most common reasons for referral to mental healthcare among children and adolescents (Antshel, 2015; Polanczyk et al., 2015). When left untreated, problems may exacerbate and put children at risk of adverse outcomes later on in life, such as school dropout, delinquency, substance use and depression (Franke et al., 2018; Reef et al., 2011). Ideally, treatment should prevent this escalation of problems, reduce the need for long and intensive treatments, and lower societal costs (Drummond et al., 2015).

   Behavioral parent training is the first psychosocial treatment of choice for reducing behavioral difficulties in preschool and school aged children (Akwa GGZ, 2019; Brestan & Eyberg, 1998; Eyberg et al., 2008; Kaminski & Claussen, 2017; National Institute for Health and Care Excellence [NICE], 2017; National Institute for Health and Care Excellence [NICE], 2019; Nederlandse Vereniging voor Psychiatrie, 2013). However, its use in clinical practice is limited by a scarcity of certified therapists, long waiting lists, and the typically long and sometimes perceived as rigid nature of behavioral parent training programs, which may lead to parents not starting or finishing behavioral parent training (Chacko et al., 2016; Evans et al., 2018; Weisenmuller & Hilton, 2021).

   To reduce these barriers, this study evaluates a brief and individually tailored behavioral parent training program for children with behavioral difficulties (the "PAINT-GGZ" program, developed by the Psychosocial ADHD & disruptive behavior INTerventions [PAINT] consortium). The brief training includes optional booster sessions for families who need additional support. The trial will generate knowledge on the (cost)effectiveness of brief parent training with optional booster sessions for children with behavioral difficulties. Brief programs are scarce, mostly do not provide booster sessions, and are mainly evaluated in prevention settings (Kolko & Lindheim, 2014; Tully & Hunt, 2015). This project fills these knowledge gaps.
2. OBJECTIVES

   The first objective of this study is to examine the short- and longer-term (i.e., one year) effectiveness of the brief and individually tailored behavioral parent training program with optional booster sessions compared to care as usual (CAU) on daily measured child behavioral difficulties (primary outcome) and on a range of secondary outcomes (see Outcomes). Additionally, we will explore whether a number of general demographic and clinical characteristics, parental attachment, parental psychopathology, parental reward responsivity, and reward and punishment sensitivity of the child moderate the short- and longer-term intervention effects on our primary outcome. The second objective is to investigate the cost-effectiveness of the program compared to CAU. As we assess cost-effectiveness based on measures at baseline and one year after the intervention, we can only draw conclusions about the cost-effectiveness on the longer term.
3. STUDY DESIGN AND SETTING

   In this two-arm multi-center randomized controlled trial, parents of children who experience behavioral difficulties in the home setting and were referred to a child mental healthcare center, are randomly assigned (1:1 ratio) to either (a) three sessions of brief behavioral parent training with optional booster sessions, or (b) CAU, as regularly provided by the involved mental healthcare centers. There are no restrictions regarding the type (e.g., psychoeducation, parent counseling and support, individual child therapy, medication) or duration of CAU, only the brief parent training investigated in this trial is not allowed. Both parents and children in the brief behavioral parent training group are not allowed to receive CAU until the first posttreatment assessment (T1). After that, CAU is allowed and parents can also make use of booster sessions with the therapist who provided the training.

   To ensure our findings reflect the real-world impact of brief behavioral parent training (i.e., to test effectiveness rather than efficacy), the trial is fully embedded in routine mental healthcare. The participating centers are academic and non-academic youth mental healthcare centers of various sizes. Therapists who provide the brief behavioral parent training have a master's degree in psychology or child, family and education studies and have had postmaster education in cognitive behavioral therapy (at least 50 hours) or have a registered higher vocational education degree as social worker in cognitive behavioral therapy. The therapists are trained in the brief parent training by supervisors qualified in cognitive behavior therapy during a one-day training of seven hours, in which therapists practice the parent training by roleplay and evaluate on their performance. Therapists also receive weekly supervision by these qualified supervisors when providing the brief parent training. Additionally, the supervisors provide feedback to each therapist on the audio-taped first session regarding protocol fidelity, intervention integrity, and the process of providing the training (e.g., engaging parents, didactic skills). There are no in- or exclusion criteria for clinicians in the CAU condition. To prevent contamination of the two research arms, therapists never provide both the brief behavioral parent training and CAU to parents participating in this study and are instructed not to share information about the contents of the brief training.
4. TIME FRAME

   Year 1: start recruitment, screening and inclusion of parents and children, start running interventions Years 2-4: ongoing contacts with mental health care organizations; recruitment, screening, and inclusion of children; run interventions and conduct measurements; supervision of therapists; fidelity checks; other project management activities; data-analysis. The last inclusion of patients is planned in year 4.

   Year 5: further data-analysis, dissemination of results, implementation activities.

   For this trial we have installed a parent advisory board (four members, one of them represents "Balans", a Dutch association for parents of children with developmental problems). The board is involved in this trial since the grant application. They provided feedback and ideas for the current project and meet biannually in the first and last year of the project and annually in years two, three, and four. In the last year, they will be asked to give their ideas about the interpretation of the results. The members of the board receive reimbursements for all meetings.
5. STUDY POPULATION

   The sample will consist of parents of children (2-12) with behavioral difficulties who have been referred to one of the participating Dutch mental healthcare centers. Based on our previous study that found medium-sized short term effects on daily ratings of behavioral difficulties compared to waitlist (range of Cohen's d = .35 to d = .66, Hornstra et al., 2021) and studies showing medium-sized parenting intervention effects on behavioral difficulties using parent-report rating scales (Bakker et al., 2017; Daley et al., 2014; McCart et al., 2006; Van Aar et al., 2017; Van den Hoofdakker et al., 2007), we estimate the effect of our brief behavioral parent training program as compared to CAU to be at least small (d = .25).

   A power analysis has been performed using G*Power software (Faul et al., 2007). Based on an effect size of d = .25 (f = .125), two groups and three repeated measures (T0, T1, T2 for short term effectiveness), with r = .60 between-measurement relation, a power of .80 and α = 0.05, we need at least 42 participants per group, resulting in a total of 84 participants. Given that the data are clustered, we increased the sample size with 10% (Twisk, 2010), resulting in a total of 93 participants. This is in line with the number of participants in similar studies comparing behavioral treatments to CAU (e.g., Van den Hoofdakker et al., 2007).
6. TREATMENT OF SUBJECTS

   During a period of one year, parents in the parent training condition will participate in a brief three-session parent training program with optional additional booster sessions and/or CAU after the parent training. The first two sessions will take 120 minutes and the third session will take one hour. These three sessions will be planned in three to four consecutive weeks. In between sessions, parents are asked to read some materials and practice the behavioral techniques they have learned with their child at home. After the brief parent training program, care as usual and/or additional booster sessions can be requested if deemed necessary by the parents or therapist. The additional booster sessions will take one hour each and can be requested maximally once every four weeks up to one year after the brief parent training program.

   The individual, three-session parent training program uses the behavioral techniques that were identified as effective for behavioral difficulties in our microtrial (Hornstra et al., 2021) and the broader literature (Kaminski et al., 2008; Leijten et al., 2019; Leijten et al., 2021). The program combines the stimulus control and contingency management techniques that, separately, reduced behavioral difficulties in the previous microtrial. Importantly, using functional analyses, the techniques are tailored to the specific problem behaviors that individual parents experience with their child. This individualized approach perfectly fits with the advice of our parent advisory board, that indicated that targeting individual parental needs is crucial for parents. To prevent relapse and reduce the need for more intensive treatments (including psychotropic medication, such as methylphenidate or antipsychotics), a booster session on maintenance training can be added at several time points (maximum once every four weeks) for parents wishing to receive additional support. Our parent advisory board considered the optional booster sessions as very important and helpful, as some parents may experience relinquishing of their parenting skills after finishing parent training, for example in stressful times (see also Furlong & McGilloway, 2014).

   Parents in the control condition will receive care as usual, which in Dutch mental health care typically consists of psychoeducation, parent counseling and support, medication, (longer) parent training programs, family therapy, and/or cognitive behavior therapy or other therapy for the child. The load imposed on these parents depends on the type of care they and/or their child receive. This usual care will also be provided to parents who do not participate in this study. The treatment in the control condition does therefore not impose any additional load compared to not participating in this study.
7. METHODS

   Parents will provide information on children's age and gender, on their own and children's ethnicity, educational background, and household composition, and on children's previous and ongoing pharmacological and non-pharmacological treatments, medical conditions, and clinical diagnoses (e.g., ADHD, oppositional defiant disorder [ODD], conduct disorder [CD]).

   PRIMARY AND SECONDARY STUDY PARAMETERS

   The primary outcome of the study is the severity of four individual target behavioral difficulties that parents want to address in the training. The secondary outcomes of the study are parent-reported behavioral difficulties, parent-reported child well-being, parent-reported parenting behaviors, masked audio records of mealtime routines to measure parent and child behavior, parent-reported parenting stress, parent-reported parenting self-efficacy, parent-reported quality of the parent-child relation, consumption and costs of mental health care and health state utility values. The investigators will furthermore explore parents' and therapists' evaluations of the brief parent training program. All outcomes are described in more detail below.

   MODERATORS

   In addition to the general demographic and clinical characteristics and some baseline characteristics such as the severity of behavioral problems, the candidate moderators of the study are parental attachment as measured with the 12-item version of the Revised Experiences in Close Relationship (ECR-R) questionnaire (Wei et al., 2007), parental psychopathology as measured with the 25 items of the Strengths and Difficulties questionnaire (SDQ) for parents (https://www.sdqinfo.org/Adult/), parental reward responsivity as measured with the 8-item Reward Responsiveness (RR) questionnaire (Van den Berg et al., 2010), and parent-reported child reward responsivity and punishment sensitivity as measured with 22 items of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for Children (SPSRQ-C) (Luman et al., 2012).

   STUDY PROCEDURES

   Parents of children with behavioral difficulties problems who have been referred to one of the participating Dutch mental healthcare centers will be recruited by clinicians within these centers. After the diagnostic assessment of their child and before any treatment has started, the clinicians involved in the diagnostic phase will inform parents about the study and hand out the information letter. Parents who are interested can give their contact information to the clinicians. The researchers will use this contact information to further inform parents about the research through telephone calls. If parents want to participate, the researchers will ask them to provide informed consent. Both legal caretakers (if present) of the child are asked to provide consent. Parents will have at least 14 days to decide upon participation and ask the researchers any questions. If needed, parents can ask for more time to decide upon participation. Parents can leave the study at any time for any reason if they wish to do so without any consequences.

   To measure the primary and secondary outcomes and candidate moderators of treatment response, parents in both treatment arms will be asked to make audiotapes of their mealtime routines, fill out questionnaires, and answer short daily phone calls (five days in a row) on four measurement occasions. Completing the questionnaires (including those measuring moderator variables) takes 30 to 45 minutes per measurement occasion, making the audiotapes takes about 30 minutes per measurement occasion (i.e., two recordings of 15 minutes each), and making the phone calls takes two to three minutes each. Furthermore, parents in the behavioral parent training arm fill out the ECBI-I questionnaire at the beginning of and two weeks after each booster session, which takes a couple of minutes.

   The measurements take place at baseline before randomization (T0), one week after the third session for parents in the brief behavioral parent training arm and eight weeks after T0 for parents in the CAU arm (first posttreatment measurement, T1), six months after T1 (second posttreatment measurement, T2) and twelve months after T1 (third posttreatment measurement, T3).
8. STATISTICAL ANALYSIS

   Data will be analyzed on an intention-to-treat basis. To examine the effects of the intervention on the primary and secondary outcomes, we will conduct multilevel analyses (mixed modeling), taking missing data into account (Twisk et al., 2013). Depending on the fit of the models, up to four hierarchical levels will be distinguished: outcomes (level 1), nested within children (level 2), nested within therapists (level 3), nested within healthcare centers (level 4). Random intercepts at the subject level, therapist level and healthcare center level will be included only if the Likelihood Ratio Test shows a significant improvement of the model fit. Time will be included as short-term (T1) and longer-term (T2, T3) within-subjects factors and condition (brief parent training vs. CAU) as between-subjects factor. The interaction between time and condition will be examined to interpret changes over time between conditions. To examine whether the candidate moderator variables moderate the intervention effects, these variables will also be added as interaction effects to the multilevel analyses.

   To assess the cost-effectiveness of the brief behavioral parent training compared to CAU, we will calculate the Incremental Cost Effectiveness Ratio (ICER) from a societal perspective. We will perform both a cost-utility analysis (based on QALYs) and cost-effectiveness analyses (based on the daily ratings of behavioral difficulties and based on ECBI-I scores). An ICER is calculated by dividing the difference in the total costs by the difference in the total effect (either QALYs or the daily ratings of behavioral difficulties and ECBI-I scores, respectively). In these analyses, the costs of healthcare will be used and interpolated to the previous 12 months. We will compare each ICER based on relevant willingness to pay thresholds. Bootstrapping will be used to calculate the reliability of our estimates.
9. ETHICAL CONSIDERATIONS

   Parents in the parent training condition will receive a brief parent training program that uses the behavioral techniques that were identified as effective for behavioral difficulties in our recent microtrial (Hornstra et al., 2021) and the broader literature. The risk of any physical or mental harm of the study is very low and not to be expected higher than what may be expected in daily life of the parents and their children. We will exclusively use conventional methods and interventions and the study is embedded in mental healthcare settings. The children of participating parents have been referred for behavioral difficulties and parents who visit the participating clinical institutions seek treatment for these problems. Adverse reactions of the parent training will be monitored (Allan & Chacko, 2018; Linden, 2013). After the parent training, parents wishing to receive additional guidance can request extra booster sessions and/or care as usual, depending on their needs. Tailoring the care that will be provided to parents' needs will minimize the chance of any physical or mental harm.

   The children with behavioral difficulties (i.e., minors) will not be directly involved in the study. Specifically, they will not be present during the brief parent training sessions and all measures will be parental measures. Furthermore, diverse populations and participants will not be denied treatment. To debrief participants, after the study is finished parents who wish to learn about the results of the study can request this information from the researchers. We inform parents about the possibility to ask for this information in the information letter.
10. ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION

HANDLING AND STORAGE OF DATA AND DOCUMENTS

Digital data, both raw and processed data are stored at a study specific secured folder within the network of Accare, the institution at which the research is carried out. This study specific folder can only be accessed by authorized personnel, who are involved in this study. All questionnaire data and processed audio files are stored in one, pseudonymized file, that is accompanied by a 'readme' text file that contains a code book explaining the meaning of all variables. A separate logbook-file will be created documenting all decisions that are made during the process from raw to processed data. Raw data containing identifiable information is kept strictly separate from the processed data and can only be accessed by two of the supervisors (BJvdH., TJD), research assistants and PhD candidate (RSvD). After the research project will be completed (i.e., data collection, data analysis and publishing of research articles), all digital data will be transferred to a study specific folder for long-term storage. The folder can only be accessed by authorized personnel. All research data will be stored for at least 15 years after the data collection has been completed. Upon request, the processed, pseudonymized data will be available for fellow researchers and made available (restricted access) for use in future research projects, to which all participants have consented before enrolling in the study. Requests for re-use of data will be evaluated to check whether the research question falls within the scope of the informed consent.

MONITORING AND QUALITY ASSURANCE

Intervention fidelity (i.e., the percentage of items covered in each session) is assessed with a fidelity checklist using an adapted version of the procedures of Abikoff and colleagues (Abikoff et al., 2013; Abikoff et al., 2015). This implies that all intervention sessions (including the booster sessions) are audiotaped. The audiotapes of 20% randomly selected sessions will be scored on intervention fidelity by independent evaluators. After each session, therapists also have to complete a fidelity checklist in which they are asked which items they covered.

Therapists also receive weekly supervision by these qualified supervisors when providing the brief parent training. Additionally, the supervisors provide feedback to each therapist on the audio-taped first session regarding protocol fidelity, intervention integrity, and the process of providing the training (e.g., engaging parents, didactic skills).

ELIGIBILITY:
Inclusion Criteria:

* The child is aged between 2 and 12 years;
* Parents have to identify at least four behavioral difficulties of the child that occur in the home setting and that they want to target in the training, using an adapted version of a list of target behaviors (Van den Hoofdakker et al., 2007; Hornstra et al., 2021). This list contains 29 behaviors that can be targeted in the training, such as hyperactive, impulsive, inattentive, oppositional and defiant behavior. The items are derived from target problems that parents mentioned in previous behavioral parent training groups and concern child behaviors that are commonly targeted in behavioral parent training in clinical practice, confirming ecological validity (Van den Hoofdakker et al., 2007).

Exclusion Criteria:

* The child uses psychotropic medication (currently or in the month before the screening);
* The child has at any time received a diagnosis of autism spectrum disorder (ASD) in clinical practice, as (parents of) children with ASD may have different needs and therefore may require different treatments than children with behavioral difficulties without ASD;
* The child has a known IQ-score below 70, as (parents of) children with intellectual disabilities may have different needs and therefore may require different treatments than children with behavioral difficulties and typical intellectual abilities;
* Parents received behavioral parent training aimed at reducing the behavioral difficulties of the concerned child in the year prior to the start of the study;
* It is not a suitable period for the parents and/or the child to participate in the study (e.g., moving, divorce);
* The child is not living in the same household as the parent(s) who participate(s) in the trial during at least four weekdays (to ensure that our primary outcome can be reported by the same informant(s) and that parents can apply the intervention plans at home).

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in individually determined daily ratings of behavioral difficulties | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  The primary outcome is the mean severity of parents' daily ratings of four selected target behaviors in specific home situations. On the adapted version of the list of target behaviors (Van den Hoofdakker et al., 2007; Hornstra et al., 2021), parents indicate whether the 29 behaviors occur daily (yes/no). For behaviors scored as yes, parents rate the severity on a 5-point Likert scale ranging from 1 (not severe) to 5 (extremely severe). With a researcher, parents choose four daily occurring target behaviors from this list that they prefer to work on in the training. Parents also indicate in which situation these behaviors occur. For each measurement occasion, during five consecutive weekdays, short daily phone calls with parents are made to evaluate whether the four selected target behaviors occurred in the past 24 hours in the selected situation (yes/no). For each timepoint, the average score of all four behaviors on all weekdays is used as outcome measure.

SECONDARY OUTCOMES:
Change in parent-reported behavioral difficulties | A week before T0, one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), twelve months after T1 (T3), during and two weeks after each booster session for parents who receive the brief parent training.
  Change in parent-reported child disruptive behaviors is assessed with the Intensity scale of the Eyberg Child Behavior Inventory (ECBI-I) (Eyberg & Ross, 1978). The Intensity scale consists of 36-items for parents of children aged 2 to 16 and measures the frequency of specific problem behavior on a 7-point Likert scale from 1 (never) to 7 (always). The convergent and divergent validity and the reliability of the ECBI-I are well established (Abrahamse et al., 2015).
Change in child well-being | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  Change in child well-being is assessed with the Health-Related Quality of Life Questionnaire (KINDL-R) (Ravens-Sieberer & Bullinger, 1998). Parents rate their children's quality of life on 20 items regarding emotional well-being, self-esteem, family functioning, social contacts, and school, of which the total score will be used. Parents rate the items on a Likert scale ranging from 1 (never) to 5 (all the time). The KINDL-R has revealed sufficient internal consistency (α = .82) (Bullinger et al., 2008).
Change in parenting behaviors | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  Change in parenting behaviors is assessed with the Alabama Parenting Questionnaire (APQ; Shelton et al., 1996). The APQ is a 42-item parent-report measure assessing five categories of parenting practices (involvement, positive parenting, poor monitoring/supervision, inconsistent discipline, and corporal punishment), of which the total score will be used. Parents rate their parenting on a 5-point scale ranging from 1 (never) to 5 (always), with higher scores representing higher levels of the particular parenting category. The reliability and validity of the APQ are well established (Shelton et al., 1996).
Change in observed parent and child behaviors (audiotapes - masked measure) | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), and twelve months after T1 (T3)
  Change in observed parent and child behaviors is assessed with a masked measure. Parents are asked to audio record their mealtime routines for at least 15 minutes on two different weekdays. Mealtimes are notoriously busy times in family lives and thus well suited as a setting for an ecologically valid measure. The recordings of mealtime routines are a masked measure (i.e., assessors are not aware of the intervention condition), based on the method that was used by Herbert et al. (2013). Using the recordings, the following behaviors will be scored with a global coding system: parental behavior (both supportive and non-supportive parenting), child misbehavior, and emotional talk. A subsample of recordings will be double coded until sufficient interrater reliability is established.
Change in parenting stress | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  Change in parenting stress is assessed with the Parental Stress Scale (PSS; Berry & Jones, 1995). The PSS is an 18-item parent report scale that measures positive (e.g., emotional benefits) and negative (e.g., restrictions) aspects of parenting, of which the total score will be used. Parents have to agree or disagree with statements concerning parenting on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). The adequate reliability (α = .83) and validity of the PSS have been demonstrated (Berry & Jones, 1995).
Change in parenting self-efficacy | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  Change in parenting self-efficacy is measured with the subscale Efficacy of the Parenting Sense of Competence Scale (PSOC; Johnston & Mash, 1989). On the eight items of this subscale, parents rate their capability level and problem-solving ability regarding their parental role on a 6-point scale, ranging from 1 (strongly disagree) to 6 (strongly agree). The internal consistency (α = .76) of the subscale Efficacy has been established (Johnston & Mash, 1989).
Change in quality of the parent-child relation | Before the brief training/before any intervention (T0), one week after the brief training/eight weeks after T0 (T1), six months after T1 (T2), and twelve months after T1 (T3)
  Change in quality of the parent-child relation is measured with the parent version of the Parent-Child Interaction Questionnaire-Revised (PACHIQ-R; Lange et al., 2002). On 21 items, parents rate their relationship with their child on a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree), of which the total score will be used. The PACHIQ-R has been demonstrated to have high internal consistency (ranging between α = .79 and α = .93) (Lange et al., 2002).
Evaluations of the program by parents - Questionnaire | One week after the brief training/eight weeks after T0 (T1) and twelve months after T1 (T3) for parents who receive the brief parent training.
  To measure parents' satisfaction and opinion about the brief parent training, parents are asked to fill out a self-developed satisfaction questionnaire, which is based on questions of the Parent Satisfaction Questionnaire (Bearss et al., 2013), the Therapy Attitude Inventory (Eyberg, 1993; Eyberg & Johnson, 1974), and the satisfaction questionnaire that was used in Breider et al. (2019). Parents who received the brief behavioral parent training answer 13 questions about their satisfaction with the brief behavioral parent training at T1 and three questions about their satisfaction with the booster sessions (if used) at T3 on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). Parents also grade the brief behavioral parent training generally between 1 (very bad) and 10 (excellent).
Evaluations of the program by parents - Focus Groups | After the inclusion of participants in the trial is finished, which is anticipated to be at the beginning of 2025.
  To measure parents' satisfaction and opinion about the brief parent training, one or multiple focus group(s) will be organized with a small number of parents. In this focus group the new program will be qualitatively evaluated and information about feasibility and barriers and facilitators for the implementation of the training in clinical settings will be gathered.
Evaluations of the program by therapists - Questionnaire | After the trial is finished, which is anticipated to be at the beginning of 2026.
  To measure therapists' satisfaction and opinion about the brief parent training, therapists will be asked to fill in a self-developed satisfaction questionnaire, which is based on questions of the Parent Satisfaction Questionnaire (Bearss et al., 2013), the Therapy Attitude Inventory (Eyberg, 1993; Eyberg & Johnson, 1974), and the satisfaction questionnaire that was used in Breider et al. (2019). Therapists have to answer seven questions on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree) and give the brief behavioral parent training a general grade between 1 (very bad) and 10 (excellent).
Evaluations of the program by therapists - Focus Groups | After the trial is finished, which is anticipated to be at the beginning of 2026.
  To measure therapists' satisfaction and opinion about the brief parent training, one or multiple focus group(s) will be organized with a selection of therapists from different healthcare centers who provided the brief parent training and range in years of work experience and to how many families they have provided the brief behavioral parent training. In the focus group(s), important barriers and facilitators for the implementation of the program will be identified.
Change in use of health care | Before the brief training/before any intervention (T0) and twelve months after T1 (T3).
  Change in use of mental healthcare within the organization where the child is treated is measured by drawing up an inventory (based on patient records) of the type of care (brief behavioral parent training, booster sessions, CAU) that is used and the duration (in minutes) of this care between T0 and T3 in both arms. The broader use of healthcare within and outside the mental healthcare centers is assessed with the Vragenlijst Intensieve Jeugdzorg, a Dutch questionnaire on intensive youth care (Bouwmans et al., 2012). This questionnaire assesses the use of a wide variety of healthcare, along with the child's use of education, contact with judicial authorities, and losses in the productivity of parents. Parents complete this questionnaire about the use and intensity of healthcare of both the child and themselves in the past three months. Both measures of healthcare use (i.e., inventory of care and questionnaire) will be combined to obtain a complete image of all used care.
Change in costs of health care | All costs are estimated after families' participation in the study, when their healthcare use is fully measured.
  Change in healthcare costs is estimated from a societal perspective (Drummond et al., 2015). Costs of mental healthcare are estimated by multiplying the used care by the reference prices provided in the Cost Manual of the Dutch National Health Care Institute. Costs of medication are estimated by using prices provided by the Dutch National Health Care Institute (Zorginstituut Nederland, 2020). Costs in other sectors (e.g., education, justice) are estimated by using reference prices provided in the Manual Intersectoral Costs and Benefits (Drost et al., 2014).
Change in utilities | Before the brief training/before any intervention (T0) and twelve months after T1 (T3).
  Change in utilities, also called preferred health states, is assessed using quality-adjusted life years (QALYs). QALYs range between 0 and 1, where 0 represents death and 1 perfect health. QALYs are calculated based on the EuroQol-5D-5L (EQ-5D) questionnaire (EuroQol Research Foundation, 2019; Herdman et al., 2011), which parents fill out about their child. The EuroQol-5D-5L measures the child's health with five items (mobility, self-care, daily activities, pain, and anxiety/depression) on 5-level categorical scales. EQ-5D responses will be transferred into QALYs based on the Dutch EQ-5D-5L tariff for adults (Versteegh et al., 2016), as a tariff for Dutch children is not yet available. The content and face validity of the EuroQol-5D-5L are well established (Herdman et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Van den Hoofdakker, Prof. dr., Principal Investigator — Accare Child Study Center; University Medical Center Groningen; University of Groningen; Saskia Van der Oord, Prof. dr., Principal Investigator — KU Leuven
Locations (1):
- Accare, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abikoff HB, Thompson M, Laver-Bradbury C, Long N, Forehand RL, Miller Brotman L, Klein RG, Reiss P, Huo L, Sonuga-Barke E. Parent training for preschool ADHD: a randomized controlled trial of specialized and generic programs. J Child Psychol Psychiatry. 2015 Jun;56(6):618-31. doi: 10.1111/jcpp.12346. Epub 2014 Oct 16. PMID 25318650
- [Background] Abikoff H, Gallagher R, Wells KC, Murray DW, Huang L, Lu F, Petkova E. Remediating organizational functioning in children with ADHD: immediate and long-term effects from a randomized controlled trial. J Consult Clin Psychol. 2013 Feb;81(1):113-28. doi: 10.1037/a0029648. Epub 2012 Aug 13. PMID 22889336
- [Background] Allan, C., & Chacko, A. (2018). Adverse events in behavioral parent training for children with ADHD: An under-appreciated phenomenon. The ADHD Report, 26(1), 4-9. https://doi.org/10.1521/adhd.2018.26.1.4
- [Background] Bakker MJ, Greven CU, Buitelaar JK, Glennon JC. Practitioner Review: Psychological treatments for children and adolescents with conduct disorder problems - a systematic review and meta-analysis. J Child Psychol Psychiatry. 2017 Jan;58(1):4-18. doi: 10.1111/jcpp.12590. Epub 2016 Aug 8. PMID 27501434
- [Background] Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. J Autism Dev Disord. 2013 Apr;43(4):829-40. doi: 10.1007/s10803-012-1624-7. PMID 22941342
- [Background] Berry, J. O., & Jones, W. H. (1995). The parental stress scale: Initial psychometric evidence. Journal of Social and Personal Relationships, 12, 463-472. http://dx.doi.org/10.1177/0265407595123009
- [Background] Bouwmans, 2012, Handleiding vragenlijst intensieve jeugdzorg: zorggebruik en productieverlies.
- [Background] Breider S, de Bildt A, Nauta MH, Hoekstra PJ, van den Hoofdakker BJ. Self-directed or therapist-led parent training for children with attention deficit hyperactivity disorder? A randomized controlled non-inferiority pilot trial. Internet Interv. 2019 Aug 8;18:100262. doi: 10.1016/j.invent.2019.100262. eCollection 2019 Dec. PMID 31890615
- [Background] Chow, J. C., & Wehby, J. H. (2016). Associations Between Language and Problem Behavior: a Systematic Review and Correlational Meta-analysis. In Educational Psychology Review (Vol. 30, Issue 1, pp. 61-82). Springer Science and Business Media LLC. https://doi.org/10.1007/s10648-016-9385-z
- [Background] Dekkers TJ, Hornstra R, van der Oord S, Luman M, Hoekstra PJ, Groenman AP, van den Hoofdakker BJ. Meta-analysis: Which Components of Parent Training Work for Children With Attention-Deficit/Hyperactivity Disorder? J Am Acad Child Adolesc Psychiatry. 2022 Apr;61(4):478-494. doi: 10.1016/j.jaac.2021.06.015. Epub 2021 Jul 2. PMID 34224837
- [Background] Drost, R. M. W. A., Paulus, A. T. G., Ruwaard, D., & Evers, S. M. A. A. (2014). Handleiding intersectorale kosten en baten van (preventieve) interventies. Classificatie, identificatie en kostprijzen.
- [Background] Drummond et al., (2015). Methods for the economic evaluation of health care programs (Fourth edition). Oxford University Press.
- [Background] DuPaul, G. J., & Barkley, R. A. (1992). Situational Variability of Attention Problems: Psychometric Properties of the Revised Home and School Situations Questionnaires. In Journal of Clinical Child Psychology (Vol. 21, Issue 2, pp. 178-188). Informa UK Limited. https://doi.org/10.1207/s15374424jccp2102_10
- [Background] Eyberg, S. (1993). Consumer satisfaction measures for assessing parent training programs. In L. VandeCreek, S. Knapp, & T. L. Jackson (Eds.), Innovations in clinical practice: A source book, Vol. 12, pp. 377-382). Professional Resource Press/Professional Resource Exchange.
- [Background] Eyberg SM, Johnson SM. Multiple assessment of behavior modification with families: effects of contingency contracting and order of treated problems. J Consult Clin Psychol. 1974 Aug;42(4):594-606. doi: 10.1037/h0036723. No abstract available. PMID 4847264
- [Background] Eyberg, S. M., & Pincus, D. (1999). ECBI & SESBI-R: Eyberg child behavior inventory and sutter-eyberg student behavior inventory-revised: Professional manual. Lutz, Florida: Psychological Assessment Resources.
- [Background] Eyberg, S. M., & Robinson, E. A. (1983). Conduct problem behavior: Standardization of a behavioral rating. In Journal of Clinical Child Psychology (Vol. 12, Issue 3, pp. 347-354). Informa UK Limited. https://doi.org/10.1080/15374418309533155
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Franke B, Michelini G, Asherson P, Banaschewski T, Bilbow A, Buitelaar JK, Cormand B, Faraone SV, Ginsberg Y, Haavik J, Kuntsi J, Larsson H, Lesch KP, Ramos-Quiroga JA, Rethelyi JM, Ribases M, Reif A. Live fast, die young? A review on the developmental trajectories of ADHD across the lifespan. Eur Neuropsychopharmacol. 2018 Oct;28(10):1059-1088. doi: 10.1016/j.euroneuro.2018.08.001. Epub 2018 Sep 6. PMID 30195575
- [Background] Furlong M, McGilloway S. The longer term experiences of parent training: a qualitative analysis. Child Care Health Dev. 2015 Sep;41(5):687-96. doi: 10.1111/cch.12195. Epub 2014 Sep 24. PMID 25256901
- [Background] Gottschalk et al., (1969). The measurement of psychological states through the content analysis of verbal behavior. California Press.
- [Background] Herbert SD, Harvey EA, Roberts JL, Wichowski K, Lugo-Candelas CI. A randomized controlled trial of a parent training and emotion socialization program for families of hyperactive preschool-aged children. Behav Ther. 2013 Jun;44(2):302-16. doi: 10.1016/j.beth.2012.10.004. Epub 2012 Nov 10. PMID 23611079
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Hornstra R, van der Oord S, Staff AI, Hoekstra PJ, Oosterlaan J, van der Veen-Mulders L, Luman M, van den Hoofdakker BJ. Which Techniques Work in Behavioral Parent Training for Children with ADHD? A Randomized Controlled Microtrial. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):888-903. doi: 10.1080/15374416.2021.1955368. Epub 2021 Aug 23. PMID 34424102
- [Background] Johnston, C., & Mash, E. J. (1989). A Measure of Parenting Satisfaction and Efficacy. In Journal of Clinical Child Psychology (Vol. 18, Issue 2, pp. 167-175). Informa UK Limited. https://doi.org/10.1207/s15374424jccp1802_8
- [Background] Kaminski JW, Claussen AH. Evidence Base Update for Psychosocial Treatments for Disruptive Behaviors in Children. J Clin Child Adolesc Psychol. 2017 Jul-Aug;46(4):477-499. doi: 10.1080/15374416.2017.1310044. Epub 2017 May 1. PMID 28459280
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Kolko DJ, Lindhiem O. Introduction to the special series on booster sessions and long-term maintenance of treatment gains. J Abnorm Child Psychol. 2014;42(3):339-42. doi: 10.1007/s10802-013-9849-2. No abstract available. PMID 24414018
- [Background] Lange A, Evers A, Jansen H, Dolan C. PACHIQ-R: the Parent-Child Interaction Questionnaire--revised. Fam Process. 2002 Winter;41(4):709-22. doi: 10.1111/j.1545-5300.2002.00709.x. PMID 12613126
- [Background] Leijten P, Gardner F, Melendez-Torres GJ, van Aar J, Hutchings J, Schulz S, Knerr W, Overbeek G. Meta-Analyses: Key Parenting Program Components for Disruptive Child Behavior. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):180-190. doi: 10.1016/j.jaac.2018.07.900. Epub 2018 Nov 26. PMID 30738545
- [Background] Leijten P, Melendez-Torres GJ, Gardner F. Research Review: The most effective parenting program content for disruptive child behavior - a network meta-analysis. J Child Psychol Psychiatry. 2022 Feb;63(2):132-142. doi: 10.1111/jcpp.13483. Epub 2021 Jul 9. PMID 34240409
- [Background] Linden M. How to define, find and classify side effects in psychotherapy: from unwanted events to adverse treatment reactions. Clin Psychol Psychother. 2013 Jul-Aug;20(4):286-96. doi: 10.1002/cpp.1765. Epub 2012 Jan 18. PMID 22253218
- [Background] Lipszyc J, Schachar R. Inhibitory control and psychopathology: a meta-analysis of studies using the stop signal task. J Int Neuropsychol Soc. 2010 Nov;16(6):1064-76. doi: 10.1017/S1355617710000895. Epub 2010 Aug 19. PMID 20719043
- [Background] Luman M, van Meel CS, Oosterlaan J, Geurts HM. Reward and punishment sensitivity in children with ADHD: validating the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for children (SPSRQ-C). J Abnorm Child Psychol. 2012 Jan;40(1):145-57. doi: 10.1007/s10802-011-9547-x. PMID 21789519
- [Background] Marsh AA, Blair RJ. Deficits in facial affect recognition among antisocial populations: a meta-analysis. Neurosci Biobehav Rev. 2008;32(3):454-65. doi: 10.1016/j.neubiorev.2007.08.003. Epub 2007 Sep 1. PMID 17915324
- [Background] Matthys W, Vanderschuren LJ, Schutter DJ. The neurobiology of oppositional defiant disorder and conduct disorder: altered functioning in three mental domains. Dev Psychopathol. 2013 Feb;25(1):193-207. doi: 10.1017/S0954579412000272. Epub 2012 Jul 17. PMID 22800761
- [Background] McCart MR, Priester PE, Davies WH, Azen R. Differential effectiveness of behavioral parent-training and cognitive-behavioral therapy for antisocial youth: a meta-analysis. J Abnorm Child Psychol. 2006 Aug;34(4):527-43. doi: 10.1007/s10802-006-9031-1. Epub 2006 Jul 13. PMID 16838122
- [Background] McMahon, R. J., & Forehand, R. L. (2019). Helping the Noncompliant Child. In Encyclopedia of Couple and Family Therapy (pp. 1359-1364). Springer International Publishing. https://doi.org/10.1007/978-3-319-49425-8_382
- [Background] Noordermeer SDS, Luman M, Buitelaar JK, Hartman CA, Hoekstra PJ, Franke B, Faraone SV, Heslenfeld DJ, Oosterlaan J. Neurocognitive Deficits in Attention-Deficit/Hyperactivity Disorder With and Without Comorbid Oppositional Defiant Disorder. J Atten Disord. 2020 Jul;24(9):1317-1329. doi: 10.1177/1087054715606216. Epub 2015 Oct 20. PMID 26486602
- [Background] Ravens-Sieberer U, Bullinger M. Assessing health-related quality of life in chronically ill children with the German KINDL: first psychometric and content analytical results. Qual Life Res. 1998 Jul;7(5):399-407. doi: 10.1023/a:1008853819715. PMID 9691720
- [Background] Reef J, Diamantopoulou S, van Meurs I, Verhulst FC, van der Ende J. Developmental trajectories of child to adolescent externalizing behavior and adult DSM-IV disorder: results of a 24-year longitudinal study. Soc Psychiatry Psychiatr Epidemiol. 2011 Dec;46(12):1233-41. doi: 10.1007/s00127-010-0297-9. Epub 2010 Oct 10. PMID 20936464
- [Background] Schoemaker K, Mulder H, Dekovic M, Matthys W. Executive functions in preschool children with externalizing behavior problems: a meta-analysis. J Abnorm Child Psychol. 2013 Apr;41(3):457-71. doi: 10.1007/s10802-012-9684-x. PMID 23054130
- [Background] Shelton, K. K., Frick, P. J., & Wootton, J. (1996). Assessment of Parenting Practices in Families of Elementary School-Age Children. Journal of Clinical Child Psychology, 25, 317-329. https://doi.org/10.1207/s15374424jccp2503_8
- [Background] Tully, L. A., & Hunt, C. (2015). Brief Parenting Interventions for Children at Risk of Externalizing Behavior Problems: A Systematic Review. In Journal of Child and Family Studies (Vol. 25, Issue 3, pp. 705-719). Springer Science and Business Media LLC. https://doi.org/10.1007/s10826-015-0284-6
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725
- [Background] Van den Berg I, Franken IH, Muris P. A new scale for measuring reward responsiveness. Front Psychol. 2010 Dec 31;1:239. doi: 10.3389/fpsyg.2010.00239. eCollection 2010. PMID 21922010
- [Background] van den Hoofdakker BJ, van der Veen-Mulders L, Sytema S, Emmelkamp PMG, Minderaa RB, Nauta MH. Effectiveness of behavioral parent training for children with ADHD in routine clinical practice: a randomized controlled study. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1263-1271. doi: 10.1097/chi.0b013e3181354bc2. PMID 17885567
- [Background] Weeland J, van Aar J, Overbeek G. Dutch Norms for the Eyberg Child Behavior Inventory: Comparisons with other Western Countries. J Psychopathol Behav Assess. 2018;40(2):224-234. doi: 10.1007/s10862-017-9639-1. Epub 2017 Dec 2. PMID 29937620
- [Background] Wei M, Russell DW, Mallinckrodt B, Vogel DL. The Experiences in Close Relationship Scale (ECR)-short form: reliability, validity, and factor structure. J Pers Assess. 2007 Apr;88(2):187-204. doi: 10.1080/00223890701268041. PMID 17437384
- [Background] Weisenmuller C, Hilton D. Barriers to access, implementation, and utilization of parenting interventions: Considerations for research and clinical applications. Am Psychol. 2021 Jan;76(1):104-115. doi: 10.1037/amp0000613. Epub 2020 Mar 5. PMID 32134281
- [Derived] van Doornik RS, van der Oord S, Luijckx J, Groenman AP, Leijten P, Luman M, Hoekstra PJ, van den Hoofdakker BJ, Dekkers TJ. The short- and longer-term effects of brief behavioral parent training versus care as usual in children with behavioral difficulties: study protocol for a randomized controlled trial. BMC Psychiatry. 2024 Mar 12;24(1):203. doi: 10.1186/s12888-024-05649-8. PMID 38475768